CLINICAL TRIAL: NCT04047927
Title: A Single Arm, Open-label First In Human Study for Assessing the Safety and Performance of the EpiFinder in Subjects With Clinical Indication for Lumbar Epidural Steroids Injection (ESI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omeq Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCL-100-01
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EpiFinder (Experimental): Eligible subjects will be included to this group to receive an epidural injection of steroids to treat their chronic back pain. The investigational device will be used in conjugation to the standard practice of epidural injections, to assist the investigator to identify the epidural space.
  Interventions: Device: EpiFinder

INTERVENTIONS:
Device: EpiFinder — The EpiFinder is a sensing device intended to assist physicians performing placement of epidural needle analgesic and/or anesthesia injection in a safely and accurately manner. The device is a single use sterile device consisting of a probe (Stylet), an actuator (micro DC motor), IR sensor and Controller. The device is integrated to a standard LOR Syringe and an 18G Tuohy needle and enables to simultaneously work with the standard LOR technique.

SUMMARY:
The EpiFinder device, which is the investigational device in this study, is intended for use in epidural procedures, between a luer syringe and an epidural needle, to give the treating physician a clear indication that the needle tip has entered the epidural space. The objective of this First In Human study is to evaluate the safety and performance of using the EpiFinder to identify the epidural space in subjects with a clinical indication to receive a lumbar Epidural Steroid Injections.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject with clinical indication for lumbar ESI based on subject's clinical problem (e.g. DDD hernia disc, spinal stenosis)
* Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed

Exclusion Criteria:

* Subject with marked spinal deformities
* Previous back surgery
* Contraindication for epidural injections (e.g. continuous use of anticoagulants, infection, allergic reactions to the injected substances)
* Subject has known hypersensitivity to contrast media that cannot be pre-medicated
* Subject with severe obesity (body mass index >35 kg/m2)
* Subject observed seizure within 7 days prior to study enrollment
* Subject presenting for emergency
* Subject has a skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) in their lumbar region
* Subject is pregnant (to be determined by urine pregnancy test)
* Subject who is currently participating or has participated in an investigational study, within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Safety - Device Related Serious Adverse Events | 14 days
  cumulative incidence of device-related complications and Serious adverse events (AE), observed during the procedure and throughout the follow-up period. Device related adverse events include: dural puncture with or without headache, epidural hematoma, seizures, neurological deficit or relevant device complications.
  All related and non-related adverse events will be observed on a continuous basis from the baseline through the study completion.

SECONDARY OUTCOMES:
Device Efficacy - Epidural Space Identification | Procedure
  Ability of the physician to identify the epidural space using the EpiFinder. Once the device determines that the needle tip is in the epidural space, this position will then be confirmed by epidurography
Device Performance - Physician satisfaction | Procedure
  physician's overall satisfaction from the device, as measured by a completion of an internal ease of use questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Margalit, Study Chair — Sponsor GmbH
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
All subject data will be anonymized, using only subject number and initials. All source data, such as laboratory results, will be kept on site only and will not be forwarded to the sponsor. All subject personal data will not be published.